CLINICAL TRIAL: NCT06833294
Title: Pilot of New GentleFit NIV Interfaces for Size and Fit With Pediatric Patients
Brief Title: GentleFit Non-Invasive Ventilation (NIV) Interface Trial
Status: Terminated | Type: Observational
Why Stopped: The study was terminated due to feasibility challenges related to device compatibility with the intended patient population.
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 23-021144
Record Dates: First submitted 2025-01-27; First posted 2025-02-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Device Ineffective; Device Induced Injury

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Children requiring Non-Invasive Ventilation (NIV): Children with corrected gestational age ≥ 38 weeks through 3 years old weighing > 3.5kg requiring NIV.
  Interventions: Device: GentleFit Mask, GentleFit Prong, Standard of Care Interface

INTERVENTIONS:
Device: GentleFit Mask, GentleFit Prong, Standard of Care Interface — The subject will be randomized to sequence of interfaces. The subject will wear each of three NIV interfaces for 8 cumulative hours, for a total of 24 hours. Pressure achieved using each GentleFit interface will be compared to pressure achieved by standard of care interface. In the event either the GentleFit nasal mask or nasal prong does not appropriately fit the subject, a standard of care interface will be substituted.

SUMMARY:
The primary objective is to compare pressure achieved by GentleFit Non-Invasive Ventilation (NIV) nasal mask and nasal prong to standard of care interface. Secondary objectives include to monitor skin integrity, clinical parameters, and adverse events. Additionally, to evaluate clinician opinion of ease of application and overall fit of GentleFit NIV interfaces and headgear.

DETAILED DESCRIPTION:
Current NIV interfaces commercially available do not address all size and anatomical gaps present in the pediatric population. To overcome this challenge, nasal mask and nasal prong prototype interfaces have been designed to fill some of the current size gap. These interfaces, known as GentleFit NIV, need to be trialed to ensure appropriateness of design and patient tolerance for 4-8 hour application intervals, as is standard of practice for current devices on the market.

ELIGIBILITY:
Inclusion Criteria:

1. Children with corrected gestational age ≥ 38 weeks through 3 years old weighing > 3.5kg.
2. Children who are on clinically stable Non-Invasive Ventilation (NIV) settings, defined as no escalation in support in the last 6-8 hours.
3. Children whose nares, face, or head fit at least one of the GentleFit NIV interfaces.
4. Parental/guardian permission (informed consent).

Exclusion Criteria:

1. Children whose nares, face, or head do not fit the manufacturer sizing guide for nasal mask and nasal prongs.
2. Facial anomalies (e.g. cleft lip).
3. Existing skin injury present in an area where GentleFit NIV interfaces or headgear would contact skin.
4. Patient's emergent condition.

   -

Ages: 38 Weeks to 3 Years | Sex: All
Age Groups: Child
Study Population: Children with corrected gestational age ≥ 38 weeks through 3 years old weighing > 3.5kg, requiring respiratory support via NIV.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Pressure delivered by GentleFit Nasal Mask | 24 hours
  To compare pressure achieved by GentleFit Non-invasive Ventilation (NIV) nasal mask compared to standard of care interface.
  Set Peak End Expiratory Pressure (PEEP) and Peak Inspiratory Pressure (PIP) settings and delivered PEEP, PIP and Mean Airway Pressure (MAP) will be monitored over 24 hours. Data collected from the ventilator on each interface, will be compared to the same values with standard of care interface.
Pressure delivered by GentleFit Nasal Prongs | 24 hours
  To compare pressure achieved by GentleFit NIV nasal prong compared to standard of care interface.
  Set PEEP and PIP settings and delivered PEEP, PIP and Mean Airway Pressure (MAP) will be monitored over 24 hours. Data collected from the ventilator on each interface, will be compared to the same values with standard of care interface.

SECONDARY OUTCOMES:
Skin Integrity | 24 hours
  To monitor skin integrity in compliance with Respiratory Care Procedure "Non- Invasive Ventilation Interface Skin Assessment". Skin assessments will be conducted per hospital policy as standard of care and be monitored over 24 hours. When a pressure injury is present, clinicians will use a pressure injury staging system from the National Pressure Injury Advisory Panel (NPIAP) to grade severity of skin injury when indicated. Pressure injuries will be numerically staged ( Stage 1, 2, 3 or 4), if the type of tissue injured can be visualized or directly palpated. If the wound base cannot be evaluated, classify as: a) Deep Tissue Pressure Injury (DTPI) b) Unstageable. If on a mucosal membrane, document, but do not stage.
  The numerical staging system does NOT imply linear progression of pressure injuries from Stage 1 through Stage 4, nor does it imply healing from Stage 4 through Stage 1.
Usability - Ease of Use | 24 hours
  To evaluate clinician opinion of ease of use of GentleFit NIV interfaces and headgear in pediatric subjects.
  Clinicians will complete a 5 question REDCap survey on GentleFit NIV interfaces compared to standard of care interfaces the subject is using. The clinician will rate ease of use on a scale of 1-5 with 1 rating as difficult, up to 5 being easiest over 24 hours. Comment sections are provided for free text.
Usability - Overall Fit | 24 hours
  To evaluate clinician opinion of the overall fit GentleFit NIV interfaces and headgear in pediatric subjects.
  Clinicians will complete a 5 question REDCap survey on GentleFit NIV interfaces compared to standard of care interfaces the subject is using. The clinician will evaluate the overall fit and appropriate of size of headgear and interfaces with yes/no questions over 24 hours. Comment sections are provided for free text.
Clinical Parameters - Vital Sign - Oxygen Saturation | 24 hours
  To monitor and record Oxygen Saturation (SpO2), per non-invasive ventilation standard of care, over 24 hours.
Clinical Parameters - Vital Sign - Respiratory Rate | 24 hours
  To monitor and record Respiratory Rate (RR), per non-invasive ventilation standard of care, over 24 hours.
Clinical Parameters - Vital Sign - Heart Rate | 24 hours
  To monitor and record Heart Rate (HR), per non-invasive ventilation standard of care, over 24 hours.
Clinical Parameters - Vital Sign - Transcutaneous Carbon Dioxide | 24 hours
  To monitor and record Transcutaneous Carbon Dioxide (TcPCO2) when applicable, over 24 hours.
Clinical Parameters - Ventilator Values | 24 hours
  Accurate fit is assessed by ensuring that the ventilator pressures set are delivered with accuracy while preventing skin breakdown due to inaccurate fit. Ordered verses measured ventilator settings will be recorded over 24 hours.
Occurrence of Adverse Events | 24 hours
  Presence or increased frequency/severity of events that would necessitate discontinuation of an interface. The frequencies of Adverse Events (AE)s by type, body system, severity, and relationship to study interface will be summarized over 24 hours. AE incidence will be summarized along with the corresponding exact binomial 95% two-sided confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Napolitano, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No